CLINICAL TRIAL: NCT05918796
Title: Ultrasound-guided Quadratus Lumborum Block Using Bupivacaine Versus Bupivacaine - Dexamethasone as Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Comparison Between Bupivacaine and Bupivacaine- Dexamethasone QLB for Postoperative Analgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Rasha Gamal Abusinna
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
Keywords: bupivacaine; dexamethasone; quadratus lumborum block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine (Active Comparator): ultrasound guided quadratus lumborum perineural injection of 18 ml bupivacaine (0.25%) combined with 2 ml normal saline bilaterally.
  Interventions: Drug: Bupivacaine
- bupivacaine and dexamethasone (Active Comparator): ultrasound guided quadratus lumborum perineural injection of 18 ml bupivacaine (0.25%) combined with 2ml volume of dexamethasone (8mg) bilaterally.
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine — 18 ml of bupivacaine of 0.25% injected bilaterally in quadratus lumborum block
Drug: Dexamethasone — dexamethasone
  Arms: bupivacaine and dexamethasone

SUMMARY:
The objective of this study is to assess the analgesic sparing effect of adding Dexamethasone to Bupivacaine in Quadratus lumborum block in patients undergoing Laparoscopic cholecystectomy under general anesthesia.

DETAILED DESCRIPTION:
Background: The QLB is an effective analgesic technique for various abdominal wall incisions. The QLB covers T7 to L2 dermatomes by the spread of LA drugs either into the paravertebral space or in the thoracolumbar plane, through iliohypogastric and ilioinguinal nerves, A and C fiber nociceptors, mechanoreceptors and high-density network of lumbar sympathetic fibers.

Objective: To assess the analgesic sparing effect of adding Dexamethasone to Bupivacaine in Quadratus lumborum block in patients undergoing Laparoscopic cholecystectomy under general anesthesia.

Patients and Methods: Sixty patients scheduled for elective Laparoscopic cholecystectomy surgeries under general anesthesia were included in this study, they were divided into two groups. Group A (perineural dexamethasone and bupivacaine group) [n=30] Those cases will receive 2ml volume of dexamethasone (8mg) combined with 18 ml of bupivacaine of 0.25% concentration. Group B (perineural bupivacaine group) [n=30] Those cases will receive perineural 18 ml bupivacaine (0.25%) combined with 2 ml normal saline.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aging > 18 years of both sexes.
2. Patients undergoing Laparoscopic cholecystectomy surgeries (duration of operation 50-80 minutes).
3. ASA physical status classes I - II.

Exclusion Criteria:

1. Patient's refusal of procedure or participation in the study.
2. ASA classes III or above.
3. Coagulopathy and bleeding disorders.
4. Local skin infections
5. Body mass index >40kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
measuring the time interval required till the first analgesic dose | the first 24 hours
  to reach a numeric rating scale NRS Pain score ≥4

SECONDARY OUTCOMES:
total pethidine dose received | total pethidine dose received in 24 hours
  record total dose of pethidine
mean blood pressure | will be recorded 5 minutes before injection, 5 minutes after injection then every 20 minutes intra-operatively and at intervals of 1, 2, 4, 6, 12, 18 and 24 hours postoperatively.
  hemodynamics
heart rate changes | will be recorded 5 minutes before injection, 5 minutes after injection then every 20 minutes intra-operatively and at intervals of 1, 2, 4, 6, 12, 18 and 24 hours postoperatively.
  hemodynamics
Incidence of side effects | record any side effect over 24 hours
  occurrence of nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: rasha g abusinna, MD, Principal Investigator — Faculty of medicine Ain Shams University
Locations (1):
- Ain Shams University Hospital, Cairo, EL Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No